CLINICAL TRIAL: NCT00941473
Title: Effect of Epidural Steroid Injection on Bone Mineral Density In Postmenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Charles S Day, Orthopedic Surgeon, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: J90067; IRB#4569; patient care #80211089
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: To Assess the Changes in Markers of Bone Turnover Over a Six Month Period After Epidural Steroid Inject; To Assess the Changes in Bone Mineral Density
Keywords: Epidural Injection; Bone Density
MeSH Terms: interventions — Triamcinolone Acetonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Epidural Steriod Injection (Active Comparator): This study focuses on the changes in bone mineral density over time of the cohort previously described in the inclusion criteria (post-menopausal white women)
  Interventions: Drug: Triamcinilone (kenalog)

INTERVENTIONS:
Drug: Triamcinilone (kenalog) — Epidural steroid injection of 80mg of Triamcinilone.

SUMMARY:
To evaluate for the effect of corticosteroid epidural injections on bone mineral density in postmenopausal women. Candidates for the study: Post menopausal women between the ages of 55 and 80. No history of bone disease. No thyroid/parathyroid disorder. not used injected or oral steroids in the last year. No recent smoking.

The purpose is to identify any significant change in bone mineral density with the use of epidural steroid injections. This may implicate the need for patient counseling regarding this possible side effect and the possible use of preventive measures to avoid this adverse effect.

DETAILED DESCRIPTION:
Glucocorticoids reduce bone formation and increase bone loss via a variety of mechanisms. This effect has been shown to be dose-dependent. Doses as low as 10mg of Prednisone, has been shown to lower bone density over periods as short as 20 weeks, an effect which may be prevented with use of Calcium and Vitamin D. Inhaled Tramcinilone has also been shown to lead to dose-related loss of bone at the hip in premenopausal women. Clinic visits will be arranged for recruited patients at baseline and then at 3 and 6 months after the ESI and at any time for new-onset or severe back pain. During the initial visit, consent will be obtained, patient will be given details on the study design and rationale, severity and characteristics of back pain. Epidural corticosteroid injection (ESI) has been shown to decrease pain, speed return of function, and improve neurological signs in patients presenting with low back pain.

ELIGIBILITY:
Inclusion Criteria:

Patients with low back pain and have consented to ESI. Age 55 and 5 years postmenopausal Caucasian women.

Exclusion Criteria:

1. any women who doesn't meet the inclusion criteria
2. Women with history of a disease affection bone turnover
3. Women taking any drugs known to influence bone metabolism
4. Women who had smoked within the preceding year
5. Women with abnormal serum thyrotropin concentration, or high parathyroid hormone concentratons.
6. Women who had received more than two short courses (lasting 2 weeks or less) of oral or parenteral glucocorticoids in the preceding year or any oral or pareneteral or local (intraarticular, paraspinal,...) or inhaled glucocorticoids in the preceding year
7. Women diagnosed with osteoporosis (T score<=2.5) on baseline DXA or had history of osteoportic fracture.
8. Pregnant women
9. Severe scoliosis -

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Measurements will be taken at baseline and then repeated at 3,6, and 12 months after treatment. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital W. Bloomfield, West Bloomfield, Michigan, United States